CLINICAL TRIAL: NCT06756282
Title: Pacing Dependence at 1 Year Follow-up in Patients Implanted With a Pacemaker After TAVR: a Multicenter Observational Study.
Brief Title: One Year Pacing Dependency After TAVR
Acronym: PACETAVI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Biotronik France (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-09-137
Record Dates: First submitted 2024-12-31; First posted 2025-01-01 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Patients Above 18 Years; Patient Discharge; Pacing Therapy; Aortic Stenosis (Treated With TAVI)
Keywords: transcatheter aortic valve replacement (TAVR); permanent pacing; conductive disorders; pacing dependency
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Defibrillators

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who need permanent pace maker implantation after TAVR: patients with high degree conductive disorders after TAVR who required pacemaker implantation before discharge the study will evaluated pacing dependency at one year (main objective) and the profile of patients with pacing dependency (type of initial conductive disorder, clinical characteristics)
  Interventions: Procedure: Pacemaker and defibrillator

INTERVENTIONS:
Procedure: Pacemaker and defibrillator — only patients with pacemaker implantation will be evaluated in the study

SUMMARY:
Pace maker implantation after the procedure of TAVR can be estimated at 15% of patients. However, some studies have shown that the conduction disturbances after TAVR could resolve over time, and that roughly between one- and two-thirds of patients who required a permanent pace maker implantation post TAVR were not found to be dependent at subsequent follow-up. This study aims to evaluate a cohort of patients permanently implanted with a pacemaker post-TAVR for high-grade conductive disorders and to describe the prevalence of effective pacemaker stimulation at 1 year follow-up. Secondary objectives include the evaluation of the prevalence of effective stimulation 3 months after implantation of the pace maker , description of the types of conductive disorders associated with atrial and/or ventricular stimulation, description of the initial indication for pacemaker implantation, description of the characteristics of the population with or without stimulation dependency. The objective is to better rationalize indication of permanent stimulation after TAVI

DETAILED DESCRIPTION:
A number of independent predictors have been found for long-term pacemaker dependence after TAVR that included a pre-existing RBBB, first-degree atrioventricular block, left anterior hemiblock, porcelain aorta, and implantation depth of the prosthesis However, indications for definitive cardiac stimulation after TAVR remain controversial excepted in case of complete or persistent high-grade BAV. The recommendations are particularly imprecise regarding intraventricular conductive disorders (LBBB++) and AVB 1.

Regarding the potential occurrence of more serious and delayed conductive disorders, the implantation of a pacemaker can sometimes be proposed to limit the duration of hospitalization in intensive care or ECG monitoring. The pacemaker implantation rate therefore probably does not reflect the true incidence of high-grade conductive disorders after TAVI because this rate varies greatly depending on the center, the indications for definitive stimulation still remain unclear, the rapid implantation times for a conductive disorder which risks getting worse (LBBG++) in a context of ever-shorter hospitalization periods can artificially increase the number of implantations.

the main objective of our study is therefore to evaluate a cohort of patients permanently implanted post-TAVR in our center since September 2023 for high-grade conductive disorders and to describe the prevalence of effective pacemaker stimulation at 1 year follow-up. Secondary objectives include the prevalence of effective stimulation 3 months after implantation of the definitive pace maker , description of the types of conductive disorders associated with pacing dependency at follow-up, description of the initial indication for pacemaker implantation, description of the characteristics of the population with or without stimulation dependency Describe serious clinical events at 3 months and 12 months (mortality, stroke, heart failure, rehospitalization for cardiac causes, complications related to the pace maker) Describe the profile of stimulation or non-stimulus dependent patients

ELIGIBILITY:
Inclusion Criteria:

all patients who need a permanent pacemaker implantation after TAVR

Exclusion Criteria:

Patients who have already a pace maker before TAVR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have TAVR and who are considered to need permanent pacemaker implantation before hospital discharge relating to high degree, symptomatic or not, conductive disorders
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-10-13 (Estimated)

PRIMARY OUTCOMES:
pacing dependency at 1 year follow-up | 6 months
  pacing dependency is defined:
  1. escape QRS rhythm < 30 bpm
  2. High degree atrioventricular block (paroxysmal or permanent)
  3. Atrial fibrillation with escape rhythm <40/min

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25011716/
- See also: Related Info — https://eurointervention.pcronline.com/article/pacemaker-dependency-after-transcatheter-aortic-valve-implantation-incidence-predictors-and-long-term-outcomes
- See also: Related Info — https://www.portailvasculaire.fr/sites/default/files/docs/2022_esc_evaluation_cardiovasculaire_avant_chirurgie_non_cardiaque_0.pdf